CLINICAL TRIAL: NCT01027897
Title: Pharmacokinetic and Pharmacodynamic Evaluation of Doripenem in Critically Ill Trauma Patients With Sepsis at Grady Health System
Brief Title: Pharmacokinetic and Pharmacodynamic Evaluation of Doripenem in Critically Ill Trauma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00016181a; DORICPK4003 (Other: other)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Sepsis
Keywords: Pharmacokinetics; Pharmacodynamics; Doripenem; Trauma; sepsis; Trauma patients with sepsis
MeSH Terms: conditions — Sepsis; Wounds and Injuries | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doripenem group (Experimental): Patients will receive doripenem for the treatment of their infection
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — Doripenem 1 gm administered over 4 hours X 3 doses

SUMMARY:
The study hypothesis is to measure how the drug doripenem is cleared from the body of critically ill trauma patients. The investigators will measure blood drug concentrations and calculate how much the drug distributes in the body and how fast it is removed from the body. There is little information on how drugs are cleared in critically ill patients and the wrong dose of a drug could make it ineffective. The investigators will use this information to predict the most reasonable dose to treat infections effectively in these patients.

DETAILED DESCRIPTION:
Understanding the pharmacokinetic (PK)/pharmacodynamic (PD) characteristics of an antibiotic can provide insight into developing appropriate dosing regimens. It is even more imperative at the present time to maximize PK/PD parameters since there are no new novel antimicrobial agents to treat resistant gram-negative infections. This approach allows us to achieve superior PD parameters and treat bacteria that would have been resistant to standard dosing due to higher minimum inhibitory concentrations (MICs).

Doripenem exhibits time-dependent bactericidal activity and the pharmacodynamic parameter predicting clinical and bacteriologic outcomes is the percentage of the dosing interval that free drug concentrations remain above the minimum inhibitory concentration (T > MIC) of the infecting pathogen Sepsis is known to influence drug pharmacokinetics and pharmacodynamics as a result of changes in hemodynamics, capillary permeability, third spacing, acid-base status, serum proteins, and organ function. Moreover, trauma patients tend to be younger with fewer comorbidities. They are hypermetabolic and are often given aggressive fluid resuscitation resulting in increased renal clearance of drugs and a larger volume of distribution. As a consequence of these differences in PK parameters, the calculated PD parameters will likely differ resulting in sub-optimal T> MIC. For time-dependent antibacterial agents such as doripenem, the T > MIC is one of the most important pharmacodynamic parameters in predicting clinical efficacy, therefore it is imperative to evaluate the PK parameters in this particular population.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years of age or older
* Admitted to Emory surgical intensive care unit (ICU) service
* Have a diagnosis of sepsis that requires empiric antimicrobial therapy
* Obtained written informed consent from the patient or a first-degree relative if the patient is unable to give informed consent due to his/her medical condition prior to initiation of any study procedure

Exclusion Criteria:

* Surgical ICU length of stay less than 24 hours
* Acute or chronic renal dysfunction (urine output less than 0.5 mL/kg/hr or calculated creatinine clearance of less than 50 mL/min)
* Pregnancy
* Known allergy to beta-lactam antibiotics
* Non-English-speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Salomone, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from April 2010 to July 2011. All patients were admitted to the Surgical ICU during the study period
Groups:
- Doripenem Group: Patients will receive doripenem 1 gm IV over 4 hours X 3 doses for the empiric treatment of an infection
Period: Overall Study
Arm/Group | Doripenem Group
Started | 30
Completed | 28
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doripenem Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Volume of Distribution (Vd)
Description: The Volume of distribution is the calculated volume that the given amount of drug is uniformly distributed in the body to achieve a particular concentration
Time Frame: After 3rd dose of study medication
Population: Patients that completed the study and did not have atypical variations in the measurement of serum concentrations were included in the final evaluation
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Doripenem Group
Number analyzed (Participants) | 27
liters | 28.52 (16.01)

2. Primary Outcome: Clearance (CL)
Description: Clearance is the volume of drug removed from the body per unit of time (hrs).
Time Frame: After 3rd dose of study medication
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | Doripenem Group
Number analyzed (Participants) | 27
liters per hour | 16.94 (11.4)

3. Primary Outcome: Elimination Constant (ke)
Description: The elimination rate constant of a drug from the central compartment
Time Frame: after 3rd dose of study drug
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Doripenem Group
Number analyzed (Participants) | 27
per hour | 1.47 (2.24)

ADVERSE EVENTS:
Arm/Group | Doripenem Group
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doripenem Group (N=30)
Lower gastrointestinal (Gastrointestinal disorders) | 1 (1) — Not related to drug
cardiac arrest (Cardiac disorders) | 1 (1) — Not related to drug
Post operative wound (Skin and subcutaneous tissue disorders) | 1 (1) — post operative wound infection. Not related to drug
atrial fibrillation (Cardiac disorders) | 2 (2) — Not related to drug
deep vein thrombosis (Vascular disorders) | 1 (1) — Doubtful if related to drug
renal failure acute (Renal and urinary disorders) | 2 (2) — Not related to drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No